CLINICAL TRIAL: NCT00863174
Title: A Randomized, Open Label, Two Treatment, Two Period, Two Sequence, Single Dose, Crossover, Bioequivalence Study of SPARC_147709- Test and Reference, 2mg/ml (30 mg/m2 Dose) in Patients With Multiple Myeloma
Brief Title: A Bioequivalence Study of SPARC_147709 in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DOX_21_1477_09
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Bio-equivalence
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SPARC147709
  Interventions: Drug: SPARC147709
- 2 (Active Comparator): Reference147709
  Interventions: Drug: Reference147709

INTERVENTIONS:
Drug: SPARC147709 — SPARC147709 injection
  Arms: 1
Drug: Reference147709 — Reference147709 injection
  Arms: 2

SUMMARY:
Safety and bioequivalence of SPARC_147709

ELIGIBILITY:
Inclusion Criteria:

* Availability for the entire study period and willingness to adhere to protocol requirements.
* Diagnosis of multiple myeloma and eligible for receiving Doxorubicin liposome
* 18 years of age or older
* No evidence of underlying disease (except multiple myeloma)

Exclusion Criteria:

* History or presence of significant allergy or significant history of hypersensitivity or idiosyncratic reactions to doxorubicin hydrochloride
* History of cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunologic,dermatologic, musculoskeletal, neurological or psychiatric disease.
* History of smoking (≥ 10 cigarettes/day) or consumption of tobacco products (≥ 4 chews/day).
* Positive result to HIV, HCV, RPR and HBsAg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
90% confidence interval of the relative mean Cmax, AUC0-t, AUC0-∞, of the test and reference | 2 cycles

SECONDARY OUTCOMES:
Treatment Emergent Adverse Events | 2 cycles